CLINICAL TRIAL: NCT02391025
Title: Gallium-68 Citrate PET To Detect MYC Amplification in Metastatic Castrate Resistant Prostate Cancer
Brief Title: Gallium-68 Citrate PET Used in Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 145512; NCI-2017-01773 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-03-04; First posted 2015-03-18 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Prostatic Neoplasms
Keywords: Metastatic; Prostate Cancer; Castrate Resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — gallium citrate; Gallium-68; Citric Acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gallium-68 citrate, PET (Experimental): Participants will receive a single scan obtained on a single day, followed by optional tumor biopsy within 6 weeks of scan. There will be optional follow up gallium-68 citrate PET scan to assess response to treatment received outside this study that will be completed within 12 weeks of baseline scan.
  Interventions: Drug: Gallium-68 citrate; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Gallium-68 citrate — Given via IV at time of imaging
  Other Names: Gallium-68 (8^Ga) citrate; Ga-68 citrate
Procedure: Positron Emission Tomography (PET) — Imaging procedure
  Other Names: PET Scan

SUMMARY:
This is a single center, pilot, cross-sectional imaging study investigating the use of gallium-68 citrate PET in participants with metastatic castration-resistant prostate cancer who are planning to undergo a metastatic tumor biopsy on protocol NCT02432001 (CC#125519).

The study population will consist of participants with metastatic castration-resistant prostate cancer who are undergoing a metastatic tumor biopsy as part of clinical protocol NCT02432001 (CC#125519), with evidence of resistance to androgen signaling inhibition.

DETAILED DESCRIPTION:
Primary Objective:

I. To determine the association between maximum average of standard uptake value (SUVmax-ave) of target metastatic lesions on gallium-68 citrate PET with MYC amplification determined from analysis of circulating tumor DNA.

Secondary Objectives:

I. To determine the accuracy rate, sensitivity, specificity of gallium citrate PET in the detection of metastatic lesions as compared to standard staging scans including cross-sectional imaging of the abdomen/pelvis and whole body bone scan.

II. To determine the optimal dose of gallium-68 citrate and timing of scan post-injection to maximize tumor-to-background signal.

III. To characterize the safety profile of gallium-68 citrate.

Outline:

The study will involve gallium-68 PET scan obtained on a single day, followed by optional tumor biopsy within 6 weeks of gallium scan. There will be optional follow up gallium-68 citrate PET scan to assess response to treatment that will be completed within 12 weeks of baseline gallium citrate PET.

ELIGIBILITY:
Inclusion Criteria:

* Male participants with histologically confirmed prostate cancer
* Participants must have castrate levels of testosterone (< 50 ng/dL) on Luteinizing hormone-releasing hormone (LHRH) analogue or have had prior bilateral orchiectomy, with evidence of castration-resistant disease by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria
* Age 18 years or older at the time of study entry
* Minimum of at least three discrete metastatic lesions in the bone and/or soft tissue amenable to whole body Positron Emission Tomography (PET) imaging per the judgment of study radiologist

For participants who undergo optional metastatic tumor biopsy following completion of gallium citrate PET:

* Presence of one or more metastases by standard radiographic scans that is safely accessible to tumor biopsy in the judgment of treating clinician and/or Interventional Radiology

Exclusion Criteria:

* Contra-indications to MRI, including permanent pacemaker, implantable device, aneurysm clip, or severe claustrophobia (for participants planning to be imaged on PET/ Magnetic resonance imaging(MRI) scanner)
* Active infection within 14 days of study enrollment

For participants who undergo optional metastatic tumor biopsy following completion of gallium citrate PET:

* History of radiation therapy to the target metastatic lesion selected for tumor biopsy
* Contra-indication to biopsy including uncontrolled bleeding diathesis.
* Platelets >75,000/μl and prothrombin time (PT) or international normalized ratio (INR) and a partial prothrombin time (PTT) < 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Mean maximum Standardized Uptake Value (SUVmax) | Day of imaging (1 day)
  The mean and standard deviation of SUVmax of gallium-68 citrate (across all metastatic lesions per participant) will be reported.
Mean maximum Standardized Uptake Value (SUVmax-ave) | Day of imaging (1 day)
  The mean and standard deviation of SUVmax-ave of gallium-68 citrate across all participants in the study cohort will be descriptively reported.

SECONDARY OUTCOMES:
Correlation between SUVmax and MYC gene expression | Day of imaging (1 day)
  For participants who undergo optional tumor biopsy, with evaluable RNA sequencing data: Correlation between SUVmax on Gallium-68 Citrate PET and MYC gene expression level, reported as the Pearson correlation coefficient. The coefficient correlation has a value between +1 and -1, where 1 is total positive linear correlation, 0 is no linear correlation, and -1 is total negative linear correlation.
Correlation between SUVmax and transferrin receptor gene expression | Day of imaging (1 day)
  For participants who undergo optional tumor biopsy, with evaluable RNA sequencing data: Correlation between SUVmax on Gallium-68 Citrate PET and transferrin receptor gene expression level, reported as the Pearson correlation coefficient. The coefficient correlation has a value between +1 and -1, where 1 is total positive linear correlation, 0 is no linear correlation, and -1 is total negative linear correlation.
Mean SUVmax-ave percent change from baseline | Up to 12 weeks
  For participants who undergo optional follow up gallium-68 citrate PET scan, the mean percent change from baseline in SUVmax-ave will be descriptively reported.
Sensitivity of gallium-68 PET | Day of imaging (1 day)
  Using as a cut-off to define a positive lesion on gallium-68 citrate PET as a lesion with SUV at least 1.5 times higher than mediastinal blood pool, the sensitivity value of gallium-68 PET will be descriptively reported on a lesion-per-lesion basis, using as reference standard staging scans including CT or MRI of the chest/abdomen/pelvis and whole body bone scan.
Specificity of gallium-68 PET | Day of imaging (1 day)
  Using as a cut-off to define a positive lesion on gallium-68 citrate PET as a lesion with SUV at least 1.5 times higher than mediastinal blood pool, the specificity of gallium-68 PET will be descriptively reported on a lesion-per-lesion basis, using as reference standard staging scans including CT or MRI of the chest/abdomen/pelvis and whole body bone scan.
Positive predictive value (PPV) of gallium-68 PET | Day of imaging (1 day)
  Using as a cut-off to define a positive lesion on gallium-68 citrate PET as a lesion with SUV at least 1.5 times higher than mediastinal blood pool, the positive predictive value of gallium-68 PET will be descriptively reported on a lesion-per-lesion basis, using as reference standard staging scans including CT or MRI of the chest/abdomen/pelvis and whole body bone scan.
Number of participants with reported treatment-emergent adverse events | Up to 12 weeks
  The frequency and severity of adverse events following gallium-68 citrate injection will be descriptively reported, using CTCAE version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02391025/ICF_000.pdf